CLINICAL TRIAL: NCT05960526
Title: Efficacy Of Nasal Irrigation With Combination of 0.9% NaCl and Binahong Extract (Anredera Cordifolia) 2,5% In Allergic Rhinitis
Brief Title: Nasal Irrigation With Combination of 0.9% NaCl and Binahong Extract (Anredera Cordifolia) 2,5% In Allergic Rhinitis
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, Asti Widuri, Associate Professor, Gadjah Mada University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KE/FK/0419/EC/2023
Record Dates: First submitted 2023-06-22; First posted 2023-07-25 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Allergic Rhinitis; Allergic Rhinitis Due to House Dust Mite
Keywords: nasal irrigation; herbal medicine
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nasal irrigation with Saline group (Active Comparator): The patient uses nasal irrigation with saline only and then mixed with 300 ml of water. The treatment was done by tilting the head 45 degrees, then spraying 150 ml of liquid on one side and repeating it on the other. The treatment was done twice daily (morning and evening) for 14 days.
  Interventions: Drug: Isotonic saline nasal irrigation
- nasal irrigation with Saline combination with binahong extract (Experimental): The patient uses nasal irrigation with saline and combination with Binahong Extract 2,5% and then mixed with 300 ml of water. The treatment was done by tilting the head 45 degrees, then spraying 150 ml of liquid on one side and repeating it on the other. The treatment was done twice daily (morning and evening) for 14 days.
  Interventions: Drug: extract Binahong

INTERVENTIONS:
Drug: extract Binahong — Extract Binahong 2.5% as nasal irrigation solution
  Other Names: extract Anredera cordifolia
  Arms: nasal irrigation with Saline combination with binahong extract
Drug: Isotonic saline nasal irrigation — NaCl 0.9% as nasal irrigation solution
  Other Names: Saline solution
  Arms: nasal irrigation with Saline group

SUMMARY:
This randomized control trial study aims to know the effects of adding 2,5% Binahong extract on the effectiveness of NaCl 0.9% nasal irrigation in patients with allergic rhinitis. The main questions it aims to answer are:

1. How does the efficacy of Binahong Extract 2,5% with 0,9% NaCl to mRNA expression (IL-4, Il-6, IL-13, and TNF-α)?
2. How does the efficacy of Binahong Extract 2,5% with 0,9% NaCl to clinical symptoms?
3. How does the efficacy of Binahong Extract 2,5% with 0,9% NaCl to quality of life?
4. How does the efficacy of Binahong Extract 2,5% with 0,9% NaCl to physiology? Participants will use nasal irrigation two times daily for two weeks. Researchers will compare the nasal irrigation group using a combination of Binahong Extract 2,5% with the group using NaCl only to see the superior effect.

DETAILED DESCRIPTION:
Background: Nasal irrigation with NaCl 0.9% is a recommended adjuvant therapy for sinonasal diseases, including allergic rhinitis, to reduce symptoms and the use of drugs. The nasal irrigation mechanism physically cleans irritant particles adhering to the nasal mucosa, reduce inflammation by reducing the concentration of inflammatory mediators, improve mucociliary function by increasing nasal cavity fluid, humidity and repairs the mucosal epithelium. Binahong is a medicinal plant widely used to improve mucosal conditions, accelerate wound healing, and have an anti-inflammatory effect. With the addition of 2.5% Binahong extract in NaCl 0.9% solution, anti-inflammatory substances are expected to increase the effectiveness of nasal irrigation in patients with allergic rhinitis.

Objective: To know the effects of the addition 2.5% Binahong extract on the effectiveness of NaCl 0.9% nasal irrigation in patients with allergic rhinitis with the assessment of mRNA expression (IL-4, Il-6, IL-13, and TNF-α), clinical symptoms, quality of life, physiology, also to know the effectiveness analysis of intervention and side effects.

Methods: Analytical study designed in randomized control trials parallel groups, single-blind on adults subjects with allergic rhinitis. The diagnosis of AR was based on clinical symptoms of a Score for Allergic Rhinitis ≥7, supportive physical examination, and positive skin prick test result. Participants were randomly divided into two groups who were given NaCl 0.9 % nasal wash and NaCl 0.9 % nasal wash with 2.5% Binahong extract twice a day for 2 weeks. Examination of mRNA expression (IL-4, Il-6, IL-13, and TNF-α), clinical symptoms (SNOT-22), quality of life (Mini-RQLQ), physiology (nasal flow and patency, mucociliary transport time) were performed before and after treatment. The data were described, tested for normality and homogeneity, then analyzed by t-test and if significant, continued by N-Gain score analysis.

Outcome: Scientific evidence of results for the addition of 2.5% Binahong extract to NaCl 0.9% nasal irrigation on mRNA expression (IL-4, Il-6, IL-13, and TNF-α), clinical symptoms, quality of life, and physiology.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with allergic rhinitis symptoms (SFAR score ≥7) aged 18 to 65 years, male or female
2. SPT examination results are positive
3. Agree to participate in the study by filling out written informed consent

Exclusion Criteria

1. Pregnant or breastfeeding women
2. Active smoker
3. Local allergic rhinitis
4. Patients with autoimmune diseases
5. Chronic rhinosinusitis with or without nasal polyps

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-05-06 (Actual); Primary Completion 2024-09-06 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
mRNA expression (IL-4, Il-6, IL-13, and TNF-α) | Change from baseline mRNA at two weeks.
  RNA samples were obtained from the epithelial mucosa of the nasal mucosa using a cytology brush by inserting the brush and rubbing it on the superior and medial inferior concha mucosa 2-3 times in a circular and parallel motion on both the right and left nasal cavities.

SECONDARY OUTCOMES:
Clinical symptoms | Change from score baseline of clinical symptom at two weeks
  Clinical symptoms were measured using the SNOT questionnaire with 22 questions consisting of 6 choices; no problem, a very mild problem, a mild/slight problem, a moderate problem, a severe problem, a very severe problem using likert scale. Thus the minimum value of this questionnaire is 0, and the maximum is 110. The outcome data scale will be analyzed in numerical form.
Physiology | Change from score baseline of physiology at two weeks
  Physiology is measured by calculating the time required for nasal mucociliary transport to move particles to the nasopharynx, carried out by the saccharin test, which calculates the time from when saccharin is placed in the anterior third of the inferior meatus nasal until it tastes sweet. The result will be analyzed in numerical form.

CONTACTS AND LOCATIONS:
Overall Officials: Bambang Rianto, MD OHNS, Principal Investigator — Gadjah Mada University
Locations (1):
- RS PKU Muhammadiyah, Yogyakarta, DIY, Indonesia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2023-03-13): https://cdn.clinicaltrials.gov/large-docs/26/NCT05960526/Prot_ICF_000.pdf